CLINICAL TRIAL: NCT00500890
Title: A Pilot Study Evaluating the Feasibility of an Intercontinental Phase III Chemotherapy Study for Patients With Choroid Plexus Tumors
Brief Title: Treatment of Tumors of the Choroid Plexus Epithelium
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: PI has left the institution
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0398; NCI-2012-01568 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-07-11; First posted 2007-07-13 (Estimated); Results first posted 2020-02-27 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Choroid Plexus Tumors
Keywords: Choroid Plexus Tumors; Carboplatin; Cyclophosphamide; Etoposide; Vincristine; Paraplatin; Cytoxan; Neosar
MeSH Terms: conditions — Choroid Plexus Neoplasms | interventions — Carboplatin; Cyclophosphamide; Etoposide; Vincristine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Carboplatin + Etoposide + Vincristine (Experimental): Carboplatin 350 mg/m^2 by vein, Over 2 Hours x 2 Days. Etoposide 100 mg/m^2 by vein, Over 1 Hour x 5 Days. Vincristine 1.5 mg/m^2 (by vein)IV Push Over 15 Minutes On Day 5. Radiation treatment over a period of about 6 weeks.
  Interventions: Drug: Carboplatin; Drug: Etoposide; Drug: Vincristine; Radiation: Radiation Therapy
- Cyclophosphamide + Etoposide + Vincristine (Experimental): Cyclophosphamide 1 g/m^2 by vein, Over 1 Hour x 2 Days. Etoposide 100 mg/m^2 by vein, Over 1 Hour x 5 Days. Vincristine 1.5 mg/m^2 (by vein)IV Push Over 15 Minutes On Day 5. Radiation treatment over a period of about 6 weeks.
  Interventions: Drug: Cyclophosphamide; Drug: Etoposide; Drug: Vincristine; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Carboplatin — 350 mg/m^2 by vein, Over 2 Hours x 2 Days
  Other Names: Paraplatin
  Arms: Carboplatin + Etoposide + Vincristine
Drug: Cyclophosphamide — 1 g/m^2 by vein, Over 1 Hour x 2 Days
  Other Names: Cytoxan; Neosar
  Arms: Cyclophosphamide + Etoposide + Vincristine
Drug: Etoposide — 100 mg/m^2 by vein, Over 1 Hour x 5 Days
Drug: Vincristine — 1.5 mg/m^2 (by vein)IV Push Over 15 Minutes On Day 5
Radiation: Radiation Therapy — Radiation treatment over a period of about 6 weeks.
  Other Names: RT; XRT; Radiotherapy

SUMMARY:
The goal of this clinical research study is to compare carboplatin to cyclophosphamide when given with etoposide, vincristine, and radiation therapy in the treatment of choroid plexus tumors. The safety of these 2 combination therapies will also be compared.

Objectives:

OVERALL AIM:

To improve choroid plexus tumor treatment through better understanding of the tumor biology and through increased knowledge about the benefit of specific treatment elements.

Specific Objectives:

The study will have a prephase to evaluate the feasibility of the following randomized study (main phase).

Pre-Phase (completed 2005) Primary Specific Objective:

To determine the number of patients accountable per year for randomization in a worldwide study.

Secondary Specific Objective:

To measure the number of drop outs and to describe the toxicity of the chemotherapy.

Main Phase (started in 2006) Primary Specific Objective:

To compare the survival times after cyclophosphamide based treatment with the survival times after carboplatin based treatment in choroid plexus tumor patients.

Main Phase Secondary Specific Objectives:

1. To compare the resectability of choroid plexus tumors after two blocks of cyclophosphamide based treatment with the resectability after two blocks of carboplatin based treatment.
2. To compare response rates of incompletely resected choroid plexus tumors to two blocks of cyclophosphamide based treatment with the response rates after two blocks of carboplatin based treatment.
3. To determine the prognostic relevance of histological atypia and SV40 in choroid plexus tumors.

DETAILED DESCRIPTION:
Tumors of the choroid plexus epithelium are rare. Participants in this study will have surgery to remove as much of the brain tumor as possible. Taking as much of the tumor out during surgery is generally believed to have the best result for this disease. Some participants may even have a second surgery to remove more tumor if thought necessary.

After the tumor surgery, exact treatment for each participant in this study will depend on how much of the tumor is removed during surgery and the way the tumor tissue looks under a microscope. Some participants will not require additional treatment because most or all of the tumor has been taken out. Those participants will still be on study, but they will only have observation and not receive additional treatment. Those that require additional treatment will be randomly assigned (as in the toss of a coin) to one of 2 treatment groups with an equal chance of being assigned to either group.

Chemotherapy (treatment with anti-cancer drugs) will be given as part of treatment for participants whose tumors are not completely removed surgically. Participants in one group will receive carboplatin plus etoposide, vincristine, and radiation therapy . Participants in the other group will receive cyclophosphamide plus etoposide, vincristine, and radiation therapy. Among all the known drugs for cancer, etoposide, vincristine, cyclophosphamide, and platinum drugs are the most effective against brain tumors. Carboplatin will be used because fewer side effects related to hearing should occur later on. This study also uses radiation therapy after surgery for children younger than 3 years old. Normally, chemotherapy has been used to delay radiation therapy until the child was older because of concerns about side effects. This change has been made because of the poor results achieved when chemotherapy was used to delay radiation therapy.

Chemotherapy is the one and only additional treatment that participants under 3 years of age can receive in this study. After the first 2 cycles, response will be evaluated, including all exams done at screening before you continue on treatment, if needed. Further surgery will be considered after these exams. If both you and your doctor choose to consider further surgery and agree for the procedure to be the next appropriate step, you may undergo a second surgery to remove anymore remaining tumor. After the second surgery, the chemotherapy will be again continued on the same schedule for 4 more cycles. If you did not require further surgery, you will continue on with the chemotherapy as previously planned.

For participants older than 3 years of age, radiation therapy will be a part of the treatment. It will be given after the second cycle of chemotherapy. Participants will receive radiation once per day, five days per week, over a period of about 6 weeks. Most of the participants do not need to stay in the hospital during this time. This will be followed by 6 more cycles of chemotherapy. After 6 cycles of chemotherapy, further surgery will again be considered. While on radiation treatment, you will have blood (about 2 teaspoons) drawn for routine tests 2 times a week. Before and after the finish of radiation, another blood test (2-3 teaspoons) will be taken to monitor the kidney and liver function, as well as to measure levels of hormones. You will have a physical exam, and blood (about 2 teaspoons) will be drawn for routine tests before each cycle of treatment.

Participants in the carboplatin group will receive etoposide over 1 hour on Days 1-5, carboplatin over 2 hours on Days 2 and 3, and vincristine over 15 minutes on Day 5. This will be repeated every 4 weeks for 24 weeks. Each period of 4 weeks is considered 1 cycle of treatment.

Participants in the cyclophosphamide group will receive etoposide over 1 hour on Days 1-5, cyclophosphamide over 1 hour on Days 2 and 3, and vincristine over 15 minutes on Day 5. This will be repeated every 4 weeks for 6 cycles (24 weeks) of treatment. Mesna, a drug to protect the bladder from the effects of cyclophosphamide, will be given 15 minutes before each dose of cyclophosphamide.

The chemotherapy given in this study can cause your white blood cell count to be too low. White blood cells are infection-fighting cells. If the white blood cell count is low for too long, participants in both groups may be given a drug called G-CSF (filgrastim). Filgrastim is a growth factor naturally produced in the body to increase the production of white blood cells. Filgrastim will be given as a shot under the skin starting at Day 9 after starting the chemotherapy.

The total length of treatment that you can receive will be 7 months, if you are able to complete all the cycles of the additional treatment. You will be taken off study if the disease gets worse or intolerable side effects occur, and your doctor will discuss other treatment options with you.

After completing treatment, there will be follow-up visits every 3 months for the first year. Every 6 months there will still be visits with the doctor until 4 years after completing treatment. You will continue to have follow-up visits every year after that to monitor for any signs of the disease coming back, or for as long as you would agree to allow follow-up visits. At each visit, you will have routine blood tests (about 2-3 teaspoons), checking of hormone levels, measurement of growth, and a hearing test. The effects of radiation/chemotherapy on your brain function, your ability to learn, and your quality of life will be measured. You will have a MRI of the brain, all known metastatic sites, and of the spine. Your body height and body weight will be measured. About 2 teaspoons of blood will be drawn for routine tests. Your urine will be tested for the presence of blood. You will have a spinal tap to look for cancer cells in the spinal fluid. Your hormone levels will also be taken to see if there are any signs of metabolic disorder and growth deficiency. This will be done with the other blood test and will not require any more extra blood samples from you.

This is an investigational study. All of the drugs used in this study are FDA approved and are commercially available. Their use together in this study is experimental. A total of up to 100 patients will take part in this multicenter study. Up to 5 will be enrolled here at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. The reference center has confirmed the receipt of slides sent (For randomization only = form 2)
2. The postoperative imaging has been done and the result is available (for randomization only = for form 2 only)
3. Indication criteria: Choroid plexus papilloma (Gr I) with histologically confirmed metastases. (For randomization only = use form 2).
4. Indication criteria: Atypical choroid plexus papilloma or anaplastic choroid plexus papilloma histology with either metastases or postoperative residual tumor. (For randomization only = use form 2).
5. Indication criteria: Choroid plexus carcinoma, regardless of histologically confirmed metastases or residual tumor. (For randomization only = use form 2).
6. Informed consent signed (required for registration = form 1, and for randomization = form 2)
7. Patients must have the following: WBC > 2000/ul, platelets >85 000/ul, serum creatinine in normal range, pregnancy test negative, hearing loss less than 30dB at 3000 Hz.

Exclusion Criteria:

1. Previous irradiation or chemotherapy. (Exclusion from randomization only)
2. The protocol did not pass the local centre required approvals, such as the Ethics Committee or the scientific review.
3. Previous immunotherapy or antiangiogenic therapy (Exclusion from randomization only)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2005-09-02 (Actual); Primary Completion 2017-12-14 (Actual); Study Completion 2017-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael E. Rytting, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Wrede B, Hasselblatt M, Peters O, Thall PF, Kutluk T, Moghrabi A, Mahajan A, Rutkowski S, Diez B, Wang X, Pietsch T, Kortmann RD, Paulus W, Jeibmann A, Wolff JEA. Atypical choroid plexus papilloma: clinical experience in the CPT-SIOP-2000 study. J Neurooncol. 2009 Dec;95(3):383-392. doi: 10.1007/s11060-009-9936-y. Epub 2009 Jun 20. PMID 19543851
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study received IRB approval August 3, 2005 and was opened to recruitment September 2, 2005. The study remained open to recruitment until December 9, 2009. The study was terminated by the local IRB on December 14, 2017.
Period: Overall Study
Arm/Group | Carboplatin + Etoposide + Vincristine | Cyclophosphamide + Etoposide + Vincristine
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Carboplatin + Etoposide + Vincristine | Cyclophosphamide + Etoposide + Vincristine | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Main Phase (Started in 2006) Primary Specific Objective
Description: To compare the survival times after cyclophosphamide based treatment with survival times after carboplatin based treatment in chroid plexus tumors patients. For analysis, there will be no difference between death by tumor progression, treatment related (toxic) reasons or unrelated reasons.
Time Frame: After randomization until the end of the observation or the death of the patient
Population: No data were collected due to early termination.
Groups:
- Carboplatin + Etoposide + Vincristine: Study participants randomized to receive chemotherapy regimine containing Carboplatin, Etoposide and Vincristine.
- Cyclophosphamide + Etoposide + Vincristine: Study participants randomized to receive chemotherapy regimine containing Cyclophosphamide, Etoposide and Vincristine.
Arm/Group | Carboplatin + Etoposide + Vincristine | Cyclophosphamide + Etoposide + Vincristine
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Secondary Objective SV40
Description: To determine the prognostic relevance of histological atypia and SV40 in choroid plexus tumors. Prognosis of tumors with or without SV40 will be compared using overall survival time as endpoint. Kaplan Meier survival estimates and log rank tests as statistical methods similar to the analysis of primary objective.
Time Frame: No data were collected due to early termination
Population: No data were collected due to early termination
Arm/Group | Carboplatin + Etoposide + Vincristine | Cyclophosphamide + Etoposide + Vincristine
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Secondary Objective Resectability
Description: To compare the resectability of choroid plexus tumors after two blocks of cyclophosphamide based therapy treatment with the resectability after two blocks of carboplatin based treatment. Success of surgery after first 2 cycles of chemotherapy will be compared between two treatment arms. Percentage of patients with secondary complete remission from those with incomplete primary resection, will be used to analyze question. Tumor with CR and tumors which could be completely resected after two cycles of chemotherapy will be counted together. Frequency will be compared a month the 2 treatment arms using Chi-square test.
Time Frame: No data were collected due to early termination
Population: No data were collected due to early termination.
Arm/Group | Carboplatin + Etoposide + Vincristine | Cyclophosphamide + Etoposide + Vincristine
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Secondary Objective Response
Description: To compare response rates of incompletely resected choroid plexus tumors to two blocks of cyclophosphamide based therapy treatment with the response rates after two blocks of carboplatin based treatment.
Time Frame: No data were collected due to early termination
Population: No data were collected due to early termination
Arm/Group | Carboplatin + Etoposide + Vincristine | Cyclophosphamide + Etoposide + Vincristine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of first dosing of protocol defined treatment until 30 days after last dose of study treatment.
Arm/Group | Carboplatin + Etoposide + Vincristine | Cyclophosphamide + Etoposide + Vincristine
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carboplatin + Etoposide + Vincristine (N=1) | Cyclophosphamide + Etoposide + Vincristine (N=1)
Neutropenic Fever (Infections and infestations) | 0 | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2007-10-12): https://cdn.clinicaltrials.gov/large-docs/90/NCT00500890/Prot_SAP_000.pdf